CLINICAL TRIAL: NCT03971630
Title: Tele-monitoring of Patients With Home Mechanical Ventilation. "MyVENT" Study.
Brief Title: Tele-monitoring of Patients With Home Mechanical Ventilation (HMV) Trough Telemedicine System (MyVENT)
Acronym: MyVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fundació Eurecat (Other)
Responsible Party: Principal Investigator, Ferran Barbe, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyVENT1
Record Dates: First submitted 2019-05-27; First posted 2019-06-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Ventilatory Failure
Keywords: HMV; Tele-monitoring; Telemedicine; Chronic hypercapnic respiratory failure
MeSH Terms: conditions — Hypoventilation | interventions — Telemedicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care group (No Intervention): These patients will be followed by standard protocol in the Unit of HMV of the University Hospital of Santa María- University Hospital Arnau de Vilanova.
- MyVENT group (Experimental): These patients will be followed up using the telemedicine (MyVENT System and APP)
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Patients will be followed up using the MyVENT System and APP
  Arms: MyVENT group

SUMMARY:
The purpose of this study is to improve HMV treatment adherence using an integrated telemedicine platform (MyVENT system)

DETAILED DESCRIPTION:
The investigators propose a study to evaluate the effect of using tele-monitoring in the follow-up of patients with HMV in order to improve their compliance and evaluate its cost-effectiveness. Telemedicine will be provided by an integrated platform composed by a website and a smartphone application for achieve a real feedback between patients and clinicians.

Design: Prospective randomized clinical study that will include 184 patients with HMV. The study will be divided in two phases, the first one consisting on the website and App system development and the second one consisting on a clinical trial where the two follow-up systems (standard care vs MyVENT group) will be compared.

Randomization: Patients will be randomised into two groups, HMV treatment management with standard care vs. telemedicine follow up.

Intervention:

Group 1:MyVENT group: patients will be followed up by tele-monitoring support. MyVENT System will be updated with data extracted from the ventilation equipment. This information and the results of the complementary tests will be sent to the clinician.

Moreover, with MyVENT APP patients will receive information about their treatment and advices to improve therapy if needed.

Group 2: Standard care. In this group all the visits will be performed at hospital following daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over to 18 years old.
* Signed informed consent.
* Good knowledge about the use of smartphones.
* Patients with Chronic Obstructive Pulmonary Disease (COPD), obesity-hypoventilation syndrome and chest wall disorders who had started HMV at least three months before their inclusion.

Exclusion Criteria:

* Chronic pathology limiting life expectancy less than 1 year.
* Psychiatric limiting problems.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to HMV treatment. | 9 months
  The number of treatment hours will be obtained by the system counter

SECONDARY OUTCOMES:
Treatment efficiency | 9 months
  Reduce or maintain carbon dioxide (CO2) in the measures
Cost effectiveness | 9 months
  In both arms the evaluation of the cost effectiveness will be made at the end of the study in each group including: (telemedicine cost, HMV carrying charge, number of visits and calls).
Early detection of problems | 9 months
  In MyVENT group the system will send notices to the clinician if it detects any problem in order to solve problems earlier.
Define the patient satisfaction | 9 months
  The study will evaluate the experience of the patient in both follow-up models they will be asked about their satisfaction grade with the follow up care provided during the study using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé Illa, Principal Investigator — Spanish Respiratory Society
Locations (1):
- Hospital Universitario Arnau de Vilanova, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No